CLINICAL TRIAL: NCT04074161
Title: Effect and Safety of Subcutaneous Semaglutide 2.4 mg Once Weekly Compared to Liraglutide 3.0 mg Once Daily on Weight Management in Subjects With Overweight or Obesity
Brief Title: Research Study to Investigate How Well Semaglutide Works Compared to Liraglutide in People Living With Overweight or Obesity
Acronym: STEP 8
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9536-4576; U1111-1233-0977 (Other: World Health Organization (WHO))
Record Dates: First submitted 2019-08-28; First posted 2019-08-29 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — semaglutide; Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Semaglutide once weekly vs liraglutide once daily treatment will be open label, but each of the two active treatment arms will be double blinded against placebo administered at the same dosing frequency.
  Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Semaglutide (Experimental): Semaglutide administered s.c. (subcutaneously, under the skin) adjunct to a reduced-calorie diet and increased physical activity
  Interventions: Drug: Semaglutide
- Placebo (semaglutide) (Placebo Comparator): Placebo (semaglutide) administered s.c. adjunct to a reduced-calorie diet and increased physical activity
  Interventions: Drug: Placebo (semaglutide)
- Liraglutide (Active Comparator): Liraglutide administered s.c. adjunct to a reduced-calorie diet and increased physical activity
  Interventions: Drug: Liraglutide
- Placebo (liraglutide) (Placebo Comparator): Placebo (liraglutide) administered s.c. adjunct to a reduced-calorie diet and increased physical activity
  Interventions: Drug: Placebo (liraglutide)

INTERVENTIONS:
Drug: Semaglutide — Dose gradually increased to 2.4 mg administered once weekly for 68 weeks
  Arms: Semaglutide
Drug: Placebo (semaglutide) — Administered once weekly for 68 weeks
  Arms: Placebo (semaglutide)
Drug: Liraglutide — Dose gradually increased to 3.0 mg administered once daily for 68 weeks
  Arms: Liraglutide
Drug: Placebo (liraglutide) — Administered once daily for 68 weeks
  Arms: Placebo (liraglutide)

SUMMARY:
This study will look at participants' body weight from the start to the end of the study. The study will last for about 1½ years. This is to compare the effect on body weight in people taking semaglutide once a week or people taking liraglutide once every day. Participants will either get semaglutide, liraglutide or "dummy" medicine. Which treatment is decided by chance. Participants who receive semaglutide or semaglutide "dummy" medicine will need to take 1 injection once a week. Participants who receive liraglutide or liraglutide "dummy" medicine will need to take 1 injection once daily. The study medicine is injected with a thin needle in a skin fold in the stomach, thigh or upper arm. During the study participants will have talks with study staff about eating healthy food and how to be more physically active. Participants will have 16 clinic visits and 7 phone calls with the study doctor. At 4 of the clinic visits participants cannot eat and drink (water is allowed) for 8 hours before the visit. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older at the time of signing informed consent
* Body mass index (BMI) equal to or above 30.0 kg/m^2 or equal to or above 27.0 kg/m^2 with the presence of at least one of the following weight-related comorbidities (treated or untreated): hypertension, dyslipidaemia, obstructive sleep apnoea or cardiovascular disease
* History of at least one self-reported unsuccessful dietary effort to lose body weight

Exclusion Criteria:

* HbA1c equal to or above 48 mmol/mol (6.5%) as measured by the central laboratory at screening
* History of type 1 or type 2 diabetes mellitus
* A self-reported change in body weight of more than 5 kg (11 lbs) within 90 days before screening irrespective of medical records

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2019-09-11 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (18):
- United States (18):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Huntington Beach, California
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Plantation, Florida
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Evanston, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Baton Rouge, Louisiana
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Charleston, South Carolina
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Rockwall, Texas
  - Novo Nordisk Investigational Site, Arlington, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Result] Wharton S, Davies M, Dicker D, Lingvay I, Mosenzon O, Rubino DM, Pedersen SD. Managing the gastrointestinal side effects of GLP-1 receptor agonists in obesity: recommendations for clinical practice. Postgrad Med. 2022 Jan;134(1):14-19. doi: 10.1080/00325481.2021.2002616. Epub 2021 Nov 29. PMID 34775881
- [Result] Rubino DM, Greenway FL, Khalid U, O'Neil PM, Rosenstock J, Sorrig R, Wadden TA, Wizert A, Garvey WT; STEP 8 Investigators. Effect of Weekly Subcutaneous Semaglutide vs Daily Liraglutide on Body Weight in Adults With Overweight or Obesity Without Diabetes: The STEP 8 Randomized Clinical Trial. JAMA. 2022 Jan 11;327(2):138-150. doi: 10.1001/jama.2021.23619. PMID 35015037
- [Derived] Snitker S, Egebjerg C, Frederiksen M, Sparre T. Ease-of-use and acceptability of the novel semaglutide 2.4 mg single-dose pen-injector in people with overweight or obesity in the STEP 8 phase III trial. Diabetes Obes Metab. 2022 Nov;24(11):2273-2276. doi: 10.1111/dom.14809. Epub 2022 Aug 7. No abstract available. PMID 35791625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 19 sites in the United States (US).
Pre-assignment Details: Total 338 adults with obesity (BMI greater than or equal to (>=30.0) kilograms per square meter (kg/m^2)) or overweight (BMI >= 27.0 kg/m^2) and at least one weight-related comorbidity were randomized in a 3:1:3:1 manner to receive treatment with either semaglutide subcutaneously (s.c.) 2.4 milligram (mg) once weekly or semaglutide placebo once weekly or liraglutide s.c. 3.0 mg once daily or liraglutide placebo once daily as an adjunct to a reduced-calorie diet and increased physical activity.
Groups:
- Semaglutide 2.4 mg: The trial included an initial dose-escalation period during which the dose was gradually increased (0.24, 0.5, 1.0, 1.7 milligram (mg)) to the maintenance dose of semaglutide 2.4 mg once weekly (16-week dose-escalation period). After the dose escalation period, treatment continued on the maintenance dose up to week 68 (end of treatment). In week 44, all participants switched from the PDS290 pen-injector to the DV3396 single-dose pen-injector. A follow-up visit (end of trial) for safety assessments was scheduled 7 weeks after end of treatment.
- Liraglutide 3.0 mg: The trial included an initial dose-escalation period during which the dose was gradually increased (0.6, 1.2, 1.8, 2.4 mg) to the maintenance dose of liraglutide 3.0 mg once daily (4-week dose-escalation period). After the dose escalation period, treatment continued on the maintenance dose up to week 68 (end of treatment). A follow-up visit (end of trial) for safety assessments was scheduled 7 weeks after end of treatment.
- Pooled Placebo: Participants received placebo matched to either once weekly semaglutide or once daily liraglutide up to week 68 (end of treatment). In week 44, all participants randomized to semaglutide placebo switched from the PDS290 pen-injector to the DV3396 single-dose pen-injector. A follow-up visit (end of trial) for safety assessments was scheduled 7 weeks after end of treatment.
Period: Overall Study
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Started | 126 | 127 | 85
Full Analysis Set | 126 | 127 | 85
Safety Analysis Set | 126 | 127 | 85
Completed | 120 | 118 | 81
Not Completed | 6 | 9 | 4
Not completed — Withdrawal by Subject | 2 | 4 | 1
Not completed — Lost to Follow-up | 4 | 5 | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo | Total
Number analyzed (Participants) | 126 | 127 | 85 | 338
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48 (14) | 49 (13) | 51 (12) | 49 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 97 | 66 | 265
  Male | 24 | 30 | 19 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 7 | 39
  Not Hispanic or Latino | 111 | 110 | 78 | 299
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 94 | 95 | 60 | 249
  Race: Black or African American | 25 | 20 | 19 | 64
  Race: Asian | 4 | 6 | 3 | 13
  Race: Other | 2 | 3 | 2 | 7
  Race: Native Hawaiian or Other Pacific Islander | 1 | 3 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline (Week 0) to Week 68 in Body Weight (%) (Semaglutide 2.4 mg Versus Liraglutide 3.0 mg)
Description: Change from baseline (week 0) to week 68 in body weight (%) is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: The full analysis set (FAS) included all randomized participants. Overall Number of Participants Analyzed = participants with available data for this outcome measure. It was planned to report data only for arms 'semaglutide 2.4 mg and liraglutide 3.0 mg' for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of body weight
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg
Number analyzed (Participants) | 117 | 117
Percentage of body weight | -16.4 (10.5) | -6.4 (7.7)
Statistical Analysis 1: Comparison: Semaglutide 2.4 mg vs Liraglutide 3.0 mg; Test type: Superiority — Responses were analysed using an analysis of covariance model with randomized treatment as factor and baseline body weight as covariate; p < 0.0001, ANCOVA; Treatment difference = -9.38, 95% CI 2-sided [-11.97 to -6.80]

2. Secondary Outcome: Number of Participants Who From Baseline (Week 0) to Week 68 Achieved Body Weight Reduction Greater Than or Equal to (>=) 10% (Yes/no)
Description: Number of participants who achieved >= 10% weight reduction from baseline (week 0) to week 68 is presented. In the reported data, 'Yes' infers the number of participants who have achieved >= 10% weight reduction, whereas 'No' infers the number of participants who did not achieve >= 10% weight reduction. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to week 68
Population: FAS included all randomized participants. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 117 | 117 | 78
Participants
  Yes | 83 | 30 | 12
  No | 34 | 87 | 66

3. Secondary Outcome: Number of Participants Who From Baseline (Week 0) to Week 68 Achieved Body Weight Reduction >=15% (Yes/no)
Description: Number of participants who achieved >= 15% weight reduction from baseline (week 0) to week 68 is presented. In the reported data, 'Yes' infers the number of participants who have achieved >= 15% weight reduction, whereas 'No' infers the number of participants who did not achieve >= 15% weight reduction. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to week 68
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 117 | 117 | 78
Participants
  Yes | 65 | 14 | 5
  No | 52 | 103 | 73

4. Secondary Outcome: Number of Participants Who From Baseline (Week 0) to Week 68 Achieved Body Weight Reduction >=20% (Yes/no)
Description: Number of participants who achieved >= 20% weight reduction from baseline (week 0) to week 68 is presented. In the reported data, 'Yes' infers the number of participants who have achieved >= 20% weight reduction, whereas 'No' infers the number of participants who did not achieve >= 20% weight reduction. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: From baseline (week 0) to week 68
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 117 | 117 | 78
Participants
  Yes | 45 | 7 | 2
  No | 72 | 110 | 76

5. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Waist Circumference
Description: Change from baseline (week 0) to week 68 in waist circumference is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 114 | 113 | 76
centimeters (cm) | -13.6 (10.0) | -6.8 (8.4) | -2.0 (7.2)

6. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Body Weight (Kilograms (kg))
Description: Change from baseline (week 0) to week 68 in body weight is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 117 | 117 | 78
kilograms | -15.8 (10.2) | -6.8 (9.5) | -1.4 (9.6)

7. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Body Weight (%) (Semaglutide 2.4 mg Versus Pooled Placebo and Liraglutide 3.0 mg Versus Pooled Placebo)
Description: as for outcome 1
Time Frame: Baseline (week 0), week 68
Population: The full analysis set (FAS) included all randomized participants. Overall Number of Participants Analyzed = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage of body weight
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 117 | 117 | 78
Percentage of body weight | -16.4 (10.5) | -6.4 (7.7) | -1.6 (8.6)

8. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Systolic Blood Pressure
Description: Change from baseline (week 0) to week 68 in systolic blood pressure is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 114 | 112 | 77
millimeters of mercury (mmHg) | -7 (14) | -4 (15) | 5 (14)

9. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Diastolic Blood Pressure
Description: Change from baseline (week 0) to week 68 in diastolic blood pressure is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 114 | 112 | 77
mmHg | -5 (9) | -1 (11) | 1 (9)

10. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Total Cholesterol (Milligram Per Deciliter (mg/dL)) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in total cholesterol (measured in mg/dL) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 112 | 106 | 74
Ratio of total cholesterol | 0.92 (12.9) | 1.00 (15.0) | 0.99 (17.6)

11. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Total Cholesterol (Millimoles Per Liter (mmol/L)) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in total cholesterol (measured in mmol/L) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 112 | 106 | 76
Ratio of total cholesterol | 0.92 (12.9) | 1.00 (15.0) | 0.99 (17.6)

12. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: High Density Lipoprotein (HDL) Cholesterol (mg/dL) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in HDL cholesterol (measured in mg/dL) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 106 | 73
Ratio of HDL cholesterol | 0.99 (14.7) | 1.02 (14.4) | 0.99 (15.4)

13. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: High Density Lipoprotein (HDL) Cholesterol (mmol/L) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in HDL cholesterol (measured in mmol/L) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 106 | 73
Ratio of HDL cholesterol | 0.99 (14.7) | 1.02 (14.4) | 0.99 (15.4)

14. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Low Density Lipoprotein (LDL) Cholesterol (mg/dL) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in LDL cholesterol (measured in mg/dL) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 106 | 73
Ratio of LDL cholesterol | 0.93 (19.7) | 1.01 (23.4) | 0.99 (26.3)

15. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Low Density Lipoprotein (LDL) Cholesterol (mmol/L) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in LDL cholesterol (measured in mmol/L) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 106 | 73
Ratio of LDL cholesterol | 0.93 (19.7) | 1.01 (23.4) | 0.99 (26.3)

16. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Very Low Density Lipoprotein (VLDL) Cholesterol (mg/dL) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in VLDL cholesterol (measured in mg/dL) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 106 | 73
Ratio of VLDL cholesterol | 0.79 (33.1) | 0.89 (36.9) | 0.97 (34.7)

17. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Very Low Density Lipoprotein (VLDL) Cholesterol (mmol/L) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in VLDL cholesterol (measured in mmol/L) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 106 | 73
Ratio of VLDL cholesterol | 0.79 (33.1) | 0.89 (36.9) | 0.97 (34.7)

18. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Free Fatty Acids (FFA) (mg/dL) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in FFA (measured in mg/dL) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of FFA
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 107 | 107 | 72
Ratio of FFA | 0.90 (81.5) | 0.87 (77.7) | 1.10 (77.2)

19. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Free Fatty Acids (FFA) (mmol/L) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in FFA (measured in mmol/L) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of FFA
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 107 | 107 | 72
Ratio of FFA | 0.90 (81.5) | 0.87 (77.7) | 1.10 (77.2)

20. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Triglycerides (mg/dL) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in triglycerides (measured in mg/dL) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 106 | 73
Ratio of triglycerides | 0.80 (33.0) | 0.89 (36.7) | 0.98 (35.7)

21. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Lipids: Triglycerides (mmol/L) (Ratio to Baseline)
Description: Change from baseline (week 0) to week 68 in triglycerides (measured in mmol/L) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 106 | 73
Ratio of triglycerides | 0.80 (33.0) | 0.89 (36.7) | 0.98 (35.7)

22. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in High-sensitivity C-reactive Protein (Hs-CRP): Ratio to Baseline
Description: Change from baseline (week 0) to week 68 in hs-CRP (measured in mg/L) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of hs-CRP
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 112 | 109 | 74
Ratio of hs-CRP | 0.46 (154.1) | 0.73 (93.0) | 0.78 (71.5)

23. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Glycated Haemoglobin (HbA1c) (%)
Description: Change from baseline (week 0) to week 68 in HbA1c (%) is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percenatge of HbA1c
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 113 | 107 | 76
Percenatge of HbA1c | -0.3 (0.2) | -0.1 (0.3) | 0.1 (0.2)

24. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Glycated Haemoglobin (HbA1c) (Millimoles Per Mole (mmol/Mol))
Description: Change from baseline (week 0) to week 68 in HbA1c is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/mol
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 113 | 107 | 76
mmol/mol | -2.8 (2.6) | -1.0 (2.7) | 1.2 (2.5)

25. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Fasting Plasma Glucose (mg/dL)
Description: Change from baseline (week 0) to week 68 in fasting plasma glucose is presented. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 105 | 73
mg/dL | -9.0 (9.6) | -4.9 (10.4) | 2.4 (10.9)

26. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Fasting Plasma Glucose (mmol/L)
Description: as for outcome 25
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 111 | 105 | 73
mmol/L | -0.5 (0.5) | -0.3 (0.6) | 0.1 (0.6)

27. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Fasting Serum Insulin (Milli-international Units Per Liter (mIU/L)): Ratio to Baseline
Description: Change from baseline (week 0) to week 68 in fasting serum insulin (measured in mIU/L) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting serum insulin
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 107 | 107 | 71
Ratio of fasting serum insulin | 0.73 (57.3) | 0.85 (47.5) | 0.98 (56.8)

28. Secondary Outcome: Change From Baseline (Week 0) to Week 68 in Fasting Serum Insulin (Picomoles Per Liter (Pmol/L)): Ratio to Baseline
Description: Change from baseline (week 0) to week 68 in fasting serum insulin (measured in pmol/L) is presented as ratio to baseline. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of fasting serum insulin
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 107 | 107 | 71
Ratio of fasting serum insulin | 0.73 (57.3) | 0.85 (47.5) | 0.98 (56.8)

29. Secondary Outcome: Number of Participants at Baseline (Week 0) and Week 68 in Glycaemic Category (Normo-glycaemia, Pre-diabetes, Type 2 Diabetes (T2D))
Description: Number of participants in glycaemic categories, "normo-glycaemia, pre-diabetes and type 2 diabetes" at baseline (week 0) and 68 are presented. These categories were set as per the following criteria: 1) Normo-glycaemia: fasting plasma glucose (FPG) less than (<) 5.6 mmol/L (<100 mg/dL) and/or glycated haemoglobin (HbA1c) <5.7%; 2) Pre-diabetes: FPG 5.6 - 6.9 mmol/L (both inclusive), FPG 100 - 125 mg/dL (both inclusive) or HbA1c 5.7 - 6.4% (both inclusive); 3) Type 2 diabetes: FPG greater than or equal to (>=) 7.0 mmol/L (>=126 mg/dL) and/or HbA1c >=6.5%. Data is reported for 'in-trial' period: the uninterrupted time interval from date of randomization to date of last contact with trial site.
Time Frame: Baseline (week 0), week 68
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 110 | 111 | 77
Participants
  Baseline (week 0): normo-glycaemia | 72 | 74 | 47
  Baseline (week 0): pre-diabetes | 38 | 37 | 30
  Baseline (week 0): type 2 diabetes | 0 | 0 | 0
  Week 68: normo-glycaemia | 104 | 89 | 38
  Week 68: pre-diabetes | 5 | 21 | 36
  Week 68: type 2 diabetes | 1 | 1 | 3

30. Secondary Outcome: Number of Participants Who From Baseline (Week 0) to Week 68 Permanently Discontinued Randomized Trial Product
Description: Number of participants who from baseline (week 0) to week 68 permanently discontinued randomized trial product are presented.
Time Frame: From baseline (week 0) to week 68
Population: FAS included all randomized participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 126 | 127 | 85
Participants | 17 | 35 | 15

31. Secondary Outcome: Number of Treatment Emergent Adverse Events (TEAEs) From Baseline (Week 0) to Week 75
Description: An adverse event (AE) was any untoward medical occurrence in a clinical trial participant that was temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. All AEs mentioned here are TEAEs defined as AEs, with the onset of the event occurred in the on-treatment period. A time-point was considered on treatment if any dose of trial product has been administrated within the prior 49 days.
Time Frame: From baseline (week 0) to week 75
Population: The safety analysis set (SAS) included all randomized participants exposed to at least one dose of randomized treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 126 | 127 | 85
Events | 904 | 823 | 522

32. Secondary Outcome: Number of Serious Adverse Events (SAEs) From Baseline (Week 0) to Week 75
Description: An AE was any untoward medical occurrence in a clinical trial participant that was temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE was defined as an AE that results in death, or is life-threatening, or requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect. SAEs occurred based on the on-treatment period is presented. A time-point was considered on treatment if any dose of trial product has been administrated within the prior 49 days.
Time Frame: From baseline (week 0) to week 75
Population: SAS included all randomized participants exposed to at least one dose of randomized treatment.
Measure: Number; unit: Events
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
Number analyzed (Participants) | 126 | 127 | 85
Events | 14 | 18 | 9

ADVERSE EVENTS:
Time Frame: From week 0 to week 75
Description: All presented AEs are treatment-emergent (i.e., TEAEs). TEAEs defined as AEs, with the onset of the event occurred in the on-treatment period. Results are based on the SAS which included all randomized participants exposed to at least one dose of randomized treatment.
Arm/Group | Semaglutide 2.4 mg | Liraglutide 3.0 mg | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/127 | 0/85
Serious Adverse Events (participants affected / at risk) | 10/126 | 14/127 | 6/85
Other Adverse Events (participants affected / at risk) | 115/126 | 115/127 | 68/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=126) | Liraglutide 3.0 mg (N=127) | Pooled Placebo (N=85)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cardiac ablation (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Post procedural drainage (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Uterine enlargement (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Viral sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Semaglutide 2.4 mg (N=126) | Liraglutide 3.0 mg (N=127) | Pooled Placebo (N=85)
Abdominal distension (Gastrointestinal disorders) | 7 (9) | 9 (10) | 7 (8)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 5 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 14 (15) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (10) | 9 (10)
Bronchitis (Infections and infestations) | 5 (6) | 5 (6) | 5 (5)
COVID-19 (Infections and infestations) | 5 (5) | 11 (11) | 5 (6)
Constipation (Gastrointestinal disorders) | 49 (80) | 40 (52) | 20 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 4 (5) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 15 (15) | 16 (18) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 35 (51) | 23 (37) | 22 (26)
Dizziness (Nervous system disorders) | 10 (11) | 7 (8) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 7 (7) | 6 (7) | 5 (6)
Dyspepsia (Gastrointestinal disorders) | 11 (14) | 15 (16) | 5 (7)
Eructation (Gastrointestinal disorders) | 17 (20) | 5 (5) | 4 (4)
Fatigue (General disorders) | 12 (12) | 14 (17) | 4 (4)
Flatulence (Gastrointestinal disorders) | 10 (13) | 4 (4) | 6 (6)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (14) | 11 (13) | 5 (5)
Headache (Nervous system disorders) | 20 (46) | 18 (20) | 10 (12)
Hypertension (Vascular disorders) | 8 (8) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 14 (14) | 6 (6)
Insomnia (Psychiatric disorders) | 3 (3) | 7 (7) | 2 (2)
Nasopharyngitis (Infections and infestations) | 10 (10) | 11 (13) | 9 (11)
Nausea (Gastrointestinal disorders) | 77 (130) | 75 (102) | 19 (24)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 5 (6)
Seasonal allergy (Immune system disorders) | 1 (1) | 5 (10) | 5 (6)
Sinusitis (Infections and infestations) | 8 (9) | 8 (8) | 13 (14)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 19 (26) | 18 (23)
Urinary tract infection (Infections and infestations) | 7 (10) | 5 (5) | 2 (2)
Vomiting (Gastrointestinal disorders) | 32 (50) | 26 (34) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/61/NCT04074161/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT04074161/SAP_001.pdf